CLINICAL TRIAL: NCT02294266
Title: Mephedrone and Alcohol Interactions After Single-dose Administration in Humans
Brief Title: Mephedrone and Alcohol Interactions in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: IMIMFTCL/MEF/2
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Amphetamine-Related Disorders; Alcohol-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders; Alcohol-Related Disorders | interventions — mephedrone; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mephedrone and alcohol (Experimental): Mephedrone 200 mg, single dose, oral administration
  Alcohol 0.8g/kg diluted in lemon-flavoured water (350 ml), single dose, oral administration
  Interventions: Drug: Mephedrone and alcohol
- Mephedrone (Active Comparator): Mephedrone 200 mg, single dose, oral administration
  Lemon-flavoured water (350 ml), single dose, oral administration
  Interventions: Drug: Mephedrone
- Alcohol (Active Comparator): Lactose 200 mg, single dose, oral administration
  Alcohol 0.8g/kg diluted in lemon-flavoured water (350 ml), single dose, oral administration
  Interventions: Drug: Alcohol
- Placebo (Placebo Comparator): Lactose 200 mg, single dose, oral administration
  Lemon-flavoured water (350 ml), single dose, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mephedrone and alcohol — Single oral dose mephedrone
  Single oral dose alcohol
  Other Names: 4-methylmetcathinone; 4-MMC; Alcohol
  Arms: Mephedrone and alcohol
Drug: Mephedrone — Single oral dose mephedrone
  Other Names: 4-methylmetcathinone; 4-MMC
  Arms: Mephedrone
Drug: Alcohol — Single oral dose alcohol
  Arms: Alcohol
Drug: Placebo — Single oral dose placebo
  Other Names: Non-active treatment
  Arms: Placebo

SUMMARY:
The purposes of this study are 1) to evaluate the pharmacological effects after oral coadministration of mephedrone and alcohol and 2) determine the pharmacokinetics changes of mephedrone and alcohol concentrations after oral coadministration of mephedrone and alcohol.

DETAILED DESCRIPTION:
Mephedrone (4-methylmetcathinone, 4-MMC) is a new psychoactive substance (NPS). Mephedrone is frequently used in combination with alcohol. At present, the effects of the interaction between mephedrone and alcohol in humans have not been previously evaluated in randomized controlled clinical trials.

The aims of this study are 1) to evaluate the pharmacological effects after oral coadministration of mephedrone and alcohol and 2) determine the pharmacokinetics changes of mephedrone and alcohol concentrations after oral coadministration of mephedrone and alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent.
* Male adults volunteers (18-45 years old).
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* Recreational use of amphetamines, ecstasy and hallucinogen derivate, mephedrone or other cathinone on at least 6 occasions (two in the previous year) without any adverse reactions.
* Recreational use of alcohol (ethanol). Previous experience in acute alcohol intoxication.
* Extensive metabolizer or intermediate metabolizer phenotype for cytochrome P-450-2D6 (CYP2D6) activity determined using dextromethorphan as a selective probe drug.
* The weight does not exceed 15% of ideal weight that applies according to size and will be between 60 and 100 Kg. Minor variations will be accepted as normal limits, if the researchers considered it clinically insignificant.

Exclusion Criteria:

* Not meeting the inclusion criteria.
* Daily consumption >20 cigarettes and >4 standard units of ethanol.
* Regular use of any drug in the month prior to the study sessions. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Presence of major psychiatric disorders.
* Present history of abuse or drug dependence (except for nicotine dependence).
* Past history of drug dependence (except for nicotine dependence). Past history of drug abuse could be included.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* Blood donation 12 weeks before or participation in other clinical trials with drugs in the previous 4 weeks.
* Subjects with intolerance or serious adverse reactions to drugs or amphetamines, ecstasy and hallucinogen derivate, mephedrone or other cathinone.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Subjects with positive serology to Hepatitis B, C or HIV.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in drunkenness and drowsiness and effects | From pre-dose (baseline, 0h) to 6h post-dose
  Drunkenness and drowsiness effects will be measured using rate scales (visual analogue scales).

SECONDARY OUTCOMES:
Change in other subjective effects | From pre-dose (baseline, 0h) to 6h post-dose
  Subjective effects will be measured using rate scales (visual analogue scales, the Addiction Research Center Inventory and the Evaluation of the Subjective Effects of Substances with Abuse Potential Questionnaires). All these instruments include measures of euphoria-good effects and other feelings induced by psychostimulants and alcohol.
Change in blood pressure | From pre-dose (baseline, 0h) to 6h post-dose
  Systolic and diastolic blood pressure
Change in psychomotor function | From pre-dose (baseline, 0h) to 1, 1.5 and 4h post-dose
  Psychomotor function will be measured using Critical tracking task (CTT) and Divided Attention Task (DAT).
Change in memory function | From pre-dose (baseline, 0h) to 1, 1.5 and 4h post-dose
  Memory function will be measured using Spatial Memory Task (SMT).
Area Under the Concentration-Time Curve (AUC 0-24h) | From pre-dose (baseline, 0h) to 0.15, 0.3, 0.45, 1, 1.5, 2, 3, 4, 6, 8, and 10h post-dose
  Calculation of AUC of the concentrations of mephedrone and its metabolites in blood and urine.
Area Under the Concentration-Time Curve (AUC 0-10h) | From pre-dose (baseline, 0h) to 0.45, 1, 1.5, 2, 3, 4, 6, 8, and 10h post-dose
  Calculation of AUC of the concentrations of alcohol in blood.
Number of Participants with Serious and Non-Serious Adverse Events | 7 days after each
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators.
Elimination hal-life | From pre-dose (baseline, 0h) to 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24h post-dose
  Calculation of elimination hal-life from concentrations of mephedrone and its metabolites in blood and urine.
Elimination hal-life | From pre-dose (baseline, 0h) to 0.45, 1, 1.5, 2, 3, 4, 6, 8, an 10h post-dose
  Calculation of elimination hal-life from concentrations of alcohol in blood.
Change in heart rate | From pre-dose (baseline, 0h) to 6h post-dose
  Measure of heart rate
Change in pupil diameter | From pre-dose (baseline, 0h) to 6h post-dose
  Measure of pupil diameter
Change in oral temperature | From pre-dose (baseline, 0h) to 6h post-dose
  Measure of oral temperature

CONTACTS AND LOCATIONS:
Overall Officials: Magí Farré, MD, PhD, Principal Investigator — Institut Hospital del Mar d'Investigacions Mèdiques-IMIM. Parc
Locations (1):
- Institut Hospital del Mar d'Investigacions Mèdiques-IMIM. Parc de Salut Mar., Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Papaseit E, Perez-Mana C, de Sousa Fernandes Perna EB, Olesti E, Mateus J, Kuypers KP, Theunissen EL, Fonseca F, Torrens M, Ramaekers JG, de la Torre R, Farre M. Mephedrone and Alcohol Interactions in Humans. Front Pharmacol. 2020 Jan 28;10:1588. doi: 10.3389/fphar.2019.01588. eCollection 2019. PMID 32063845